CLINICAL TRIAL: NCT04075019
Title: The Seattle Social Development Project: A Quasi-experimental Test of the Raising Healthy Children (RHC) Intervention With Teachers, Parents, and Students in Grades 1 to 6 in Elementary Schools Serving Children From High Crime Urban Areas
Brief Title: The Seattle Social Development Project: An Implementation of the Raising Healthy Children Intervention
Acronym: SSDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, J. David Hawkins, Professor, School of Social Work, and Director, Social Development Research Group, University of Washington
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY 22-355; R01DA003721 (NIH)
Record Dates: First submitted 2019-08-27; First posted 2019-08-30 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Adolescent Health; Adolescent Problem Behavior
Keywords: Proactive classroom management; Interactive teaching; Cooperative learning; Interpersonal problem solving skills; Refusal skills; Behavior management skills; Academic support skills; Skills to reduce risks for drug use

STUDY DESIGN:
Intervention Model Description: This study examined four separate groups, a "full intervention group" exposed to the interventions in grades 1 through 6, a "late intervention group" exposed to the interventions only in grades 5 and 6, a minimal "parent-training only group" (grades 5 and 6), and a control group that received no special intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- full intervention (Experimental): students assigned to intervention classrooms in grades 1 through 4 and who remained in schools assigned to the intervention condition in grades 5 or 6
  Interventions: Behavioral: The Raising Healthy Children intervention, including teacher training, child skill development, and parent training
- late intervention (Experimental): students in intervention classrooms in grades 5 and 6 only
  Interventions: Behavioral: The Raising Healthy Children intervention, including teacher training, child skill development, and parent training
- parent-training only (Experimental): students whose parents were offered parent training only when their children were in grades 5 and 6 and no other intervention
  Interventions: Behavioral: The Raising Healthy Children intervention, including teacher training, child skill development, and parent training
- control (No Intervention): students in schools assigned to receive no intervention in grades 5 and 6 and who were not in intervention classrooms in grades 1 through 4

INTERVENTIONS:
Behavioral: The Raising Healthy Children intervention, including teacher training, child skill development, and parent training
  Other Names: Seattle Social Development Project
  Arms: full intervention; late intervention; parent-training only

SUMMARY:
The Seattle Social Development Project (SSDP) included a three-part intervention for teachers, parents, and students in grades 1 to 6. It was a universal prevention program that was tested in elementary schools serving children from high crime urban areas. The intervention trained teachers in proactive classroom management, interactive teaching, and cooperative learning. SSDP also offered training to parents in child behavior management, academic support, and skills to reduce risks for drug use. It provided training to children designed to affect interpersonal problem solving and refusal skills. These interventions were designed to reduce risks and increase protection at the individual, peer, family and school levels. The package of interventions was guided theoretically by the social development model. We hypothesized that training teachers to teach and manage their classrooms in ways that promote bonding to school, training parents to manage their families in ways that promote bonding to family and to school, and providing children with training in skills for social interaction would positively affect children's attitudes toward school, behavior at school, and academic achievement. These methods further sought to reduce children's opportunities and rewards for antisocial involvement. We thought that these changes would, in turn, set children on a different developmental trajectory observable in higher school achievement and fewer health-risk behaviors later in adolescence.

DETAILED DESCRIPTION:
The study asked whether delivering the intervention package over the full course of elementary school from grades 1 through 6 ("full intervention") had effects on academic and behavioral health outcomes; whether delivering the intervention just prior to adolescence in grades 5 and 6 only ("late intervention") had effects on academic and behavioral health outcomes; and whether offering parenting interventions only when participants were in grades 5 and 6 ("parenting only intervention") had effects on academic and behavioral health outcomes when compared with outcomes for students who were not assigned to intervention classrooms. This study examined this question by comparing outcomes for four separate groups, a "full intervention group" exposed to the interventions through grades 1-6, a "late intervention group" exposed to the interventions only in grades 5 and 6, a minimal "parent-training only group" (grades 5 and 6), and a control group that received no special intervention. The intervention package consisted of the following components:

Teacher Training In Classroom Instruction and Management included training in (a) proactive classroom management (establish consistent classroom expectations and routines at the beginning of the year; give clear, explicit instructions for behavior; recognize and reward desirable student behavior and efforts to comply; use methods that keep minor classroom disruptions from interrupting instruction); (b) interactive teaching (assess and activate foundation knowledge before teaching; teach to explicit learning objectives; model skills to be learned; frequently monitor student comprehension as material is presented; re-teach material when necessary); and (c) cooperative learning (involve small teams of students of different ability levels and backgrounds as learning partners; provide recognition to teams for academic improvement of individual members over past performance). Teacher training was provided to teachers of participants in full intervention classrooms in grades 1 through 6 and to teachers of participants in late intervention classrooms in grades 5 and 6.

Child Social and Emotional Skill Development included instruction in (a) interpersonal problem solving skills (communication; decision making; negotiation; conflict resolution) provided by teachers in classrooms assigned to the full intervention condition in grades 1 and 2; and (b) refusal skills (recognize social influences to engage in problem behaviors; identify consequences of problem behaviors; generate and suggest alternatives; invite peer(s) to join in alternatives) provided to participants in both the full intervention condition and the late intervention condition in grades 5 and 6.

Parent Training offered to parents of participants in the full intervention condition included instruction in (a) behavior management skills (observe and pinpoint desirable and undesirable child behaviors; teach expectations for behaviors; provide consistent positive reinforcement for desired behavior; provide consistent and moderate consequences for undesired behaviors) when participants were in grades 1 and 2; (b) academic support skills (initiate conversation with teachers about children's learning; help children develop reading and math skills; create a home environment supporting of learning) when participants were in grades 2 and 3; and (c) skills to reduce risks for drug use (establish a family policy on drug use; practice refusal skills with children; use self-control skills to reduce family conflict; create new opportunities in the family for children to contribute and learn) when participants were in grades 5 and 6. Parent training in skills to reduce risks for drug use was also offered to parents of participants in the late intervention condition and the parenting only condition when participants were in grades 5 and 6.

This resulted in a nonrandomized controlled trial with 4 conditions. The full intervention group received the intervention package from grade 1 through grade 6. The late intervention group received the intervention package in grades 5 and 6 only. The parent intervention only condition included students in schools assigned to receive only parent training in skills to reduce risks for drug use when their children were in grades 5 and 6, and the control group received no special intervention. This design was created in 1985 by nesting an intervention initiated in 1981 at first-grade entry within the clinical trial. For the present study, schools were assigned nonrandomly to conditions in the fall of 1985, and from that point, all fifth-grade students in the full and late intervention conditions participated in the same interventions. New schools added for the clinical trial when students entered grade 5 were matched to the original intervention and control schools with respect to grades served and inclusion of students drawn from high-crime neighborhoods of Seattle. Schools added for the panel study were assigned to conditions to achieve balanced numbers across conditions. During this study the Seattle School District used mandatory busing to achieve racial equality in schools. As a result, all schools in this study served heterogeneous population of students drawn from at least 2 different neighborhoods of the city. This practice reduced the risk that outcomes observed in the trial reflected contextual or neighborhood differences in the populations attending different schools.

ELIGIBILITY:
Inclusion Criteria:

* All students enrolled in the fifth grade in 1985 in one of 18 Seattle public elementary schools selected for the study were eligible
* Eligible schools had to serve children from neighborhoods with above average crime rates
* Parents of eligible participants consented to their longitudinal participation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 1981-09-01 (Actual); Primary Completion 1987-06-13 (Actual); Study Completion 1993-06-30 (Actual)

PRIMARY OUTCOMES:
substance use | annually at ages 10 through 16 and again at age 18 (1985 through 1991 and in 1993)
  Youth substance use was assessed by having all study participants complete standardized survey instruments from the University of Michigan Monitoring the Future survey annually from ages 10 to 16 and again at age 18, designed to assess children's substance use. Items from surveys were combined into scales assessing youth self-reported onset and use of specific substances in the year and 30 day period prior to each survey administration.
delinquency | annually at ages 10 through 16 and again at age 18 (1985 through 1991 and in 1993)
  Youth delinquency was assessed by having all study participants complete standardized survey instruments from the University of Colorado National Youth Survey annually from ages 10 to 16 and again at age 18, designed to assess children's delinquent behavior. Items from surveys were combined into scales assessing youth onset of delinquency and number of different delinquent acts self-reported by youth for the year prior to each survey administration..
school misbehavior | annually at ages 10 through 16 and again at age 18 (1985 through 1991 and in 1993)
  Youth school misbehavior was assessed by having all study participants complete standardized survey instruments annually from ages 10 to 16 and again at age 18, designed to assess children's behavioral outcomes. Teachers completed the Teacher Report Form of the Child Behavior Checklist, a standardized instrument developed to measure children's behaviors, annually from ages 11 to 14. Items from surveys were combined into scales assessing youths' self-reported onset and involvement in misbehavior at school and teacher reported involvement of the participant in misbehavior at school in the year prior to each survey administration.
aggression and violence | annually at ages 10 through 16 and again at age 18 (1985 through 1991 and in 1993)
  Youth aggression and violence was assessed by having all study participants complete standardized survey instruments annually from ages 10 to 16 and again at age 18, designed to assess children's behavioral outcomes. Teachers completed the Teacher Report Form of the Child Behavior Checklist, a standardized instrument developed to measure children's behaviors, annually from ages 11 to 14. Items from surveys were combined into scales assessing youths' self-reported onset and involvement in aggressive and violent behavior and teacher reported involvement of the participant in aggressive and violent behavior in the year prior to each survey administration.
school achievement | annually at ages 10 through 16 and again at age 18 (1985 through 1991 and in 1993)
  Youth school achievement was assessed by having all study participants complete standardized survey instruments annually from ages 10 to 16 and again at age 18, designed to assess children's behavioral outcomes. Teachers completed the Teacher Report Form of the Child Behavior Checklist, a standardized instrument developed to measure children's behaviors, annually from ages 11 to 14. Items from surveys were combined into scales assessing youths' self-reported level of achievement at school and teacher reported level of participant achievement in the year prior to each survey administration.

CONTACTS AND LOCATIONS:
Overall Officials: J. David Hawkins, PhD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: Yes
Selected, de-identified data are shared with collaborating colleagues at other institutions. Shared datasets contain variable subsets related to analyses planned for developing papers for publication.
Supporting Information: Study Protocol
Time Frame: Data first became available in 1986 and are available on an ongoing basis.
Access Criteria: Selected, de-identified data are shared with collaborating colleagues at other institutions after obtaining signed "fair use" and confidentiality agreements from the collaborator wherein they agree to work with the study PIs and abide by study-related human subjects and consent agreements, and data security procedures. Shared datasets are to be used for analyses planned for developing papers for publication. The PI is responsible for obtaining signed agreements and reviewing and approving data sharing requests.

REFERENCES:
- [Result] Hawkins JD, Von Cleve E, Catalano RF Jr. Reducing early childhood aggression: results of a primary prevention program. J Am Acad Child Adolesc Psychiatry. 1991 Mar;30(2):208-17. doi: 10.1097/00004583-199103000-00008. PMID 2016224
- [Result] Hawkins JD, Catalano RF, Morrison DM, O'Donnell J, Abbott RD, Day LE, McCord J, Tremblay RE. The Seattle Social Development Project: Effects of the first four years on protective factors and problem behaviors. In: McCord J, Tremblay, RE, editors. Preventing antisocial behavior: Interventions from birth through adolescence. New York: Guilford Press; 1992. 139-61.
- [Result] O'Donnell J, Hawkins JD, Catalano RF, Abbott RD, Day LE. Preventing school failure, drug use, and delinquency among low-income children: long-term intervention in elementary schools. Am J Orthopsychiatry. 1995 Jan;65(1):87-100. doi: 10.1037/h0079598. PMID 7733220
- [Result] Abbott RD, O'Donnell J, Hawkins JD, Hill KG, Kosterman R, Catalano RF. Changing teaching practices to promote achievement and bonding to school. Am J Orthopsychiatry. 1998 Oct;68(4):542-52. doi: 10.1037/h0080363. PMID 9809114
- [Derived] Hill KG, Steeger CM, Epstein M, Bailey JA, Hawkins JD. Addressing Suicide and Mental Health Through Universal Childhood Intervention: Results from The Seattle Social Development Project. Prev Sci. 2025 Nov;26(7):1033-1044. doi: 10.1007/s11121-025-01834-7. Epub 2025 Oct 18. PMID 41108509
- [Derived] Le VT, Bailey JA, Pandika DM, Epstein M, Satchell K. Long-term Effects of the Raising Healthy Children Intervention on Family Functioning in Adulthood: A Nonrandomized Controlled Trial. J Prev (2022). 2024 Feb;45(1):17-25. doi: 10.1007/s10935-023-00753-z. Epub 2023 Nov 16. PMID 37973659
- [Derived] Bailey JA, Pandika D, Le VT, Epstein M, Steeger CM, Hawkins JD. Testing Cross-Generational Effects of the Raising Healthy Children Intervention on Young Adult Offspring of Intervention Participants. Prev Sci. 2023 Oct;24(7):1376-1385. doi: 10.1007/s11121-023-01583-5. Epub 2023 Sep 21. PMID 37733189
- [Derived] Hill KG, Bailey JA, Steeger CM, Hawkins JD, Catalano RF, Kosterman R, Epstein M, Abbott RD. Outcomes of Childhood Preventive Intervention Across 2 Generations: A Nonrandomized Controlled Trial. JAMA Pediatr. 2020 Aug 1;174(8):764-771. doi: 10.1001/jamapediatrics.2020.1310. PMID 32511669